CLINICAL TRIAL: NCT02367456
Title: An Open-label Phase 1b Study of PF-04449913 (Glasdegib) in Combination With Azacitidine in Patients With Previously Untreated Higher-Risk Myelodysplastic Syndrome, Acute Myeloid Leukemia, or Chronic Myelomonocytic Leukemia
Brief Title: A Combination Study of PF-04449913 (Glasdegib) and Azacitidine In Untreated MDS, AML and CMML Patients
Acronym: BRIGHT 1012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1371012; 2014-001345-24 (EudraCT Number); BRIGHT MDS&AML1012 (Other: Alias Study Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: MDS; AML; CMML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — glasdegib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Arm A (Experimental): MDS patients: PF-04449913 (Glasdegib) 100 mg + Azacitidine 75 mg/m2
  Interventions: Drug: PF-04449913 (Glasdegib); Drug: Azacitidine
- Arm B (Experimental): AML patients: PF-04449913 (Glasdegib) 100 mg + Azacitidine 75 mg/m2
  Interventions: Drug: PF-04449913 (Glasdegib); Drug: Azacitidine

INTERVENTIONS:
Drug: PF-04449913 (Glasdegib) — Daily dose of PF-04449913 100mg tablet in a continuous regimen of 28 day cycles
Drug: Azacitidine — 75mg/m2 on Days 1-7 (+/- 3 days for each dose) of a 28 day cycle

SUMMARY:
This multi center open label Phase 1b study is designed to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of glasdegib (PF-04449913) when combined with azacitidine in patients with previously untreated Higher Risk Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML), or Chronic Myelomonocytic Leukemia (CMML). This clinical study includes two components: (a) a safety lead in cohort (LIC) and (b) an expansion phase with an AML cohort and an MDS cohort.

ELIGIBILITY:
Inclusion criteria:

* Patients must have previously untreated MDS, AML, or CMML according to the WHO 2016 classification.
* MDS patients must have Intermediate (>3 to 4.5 points), High Risk (>4.5 - 6) or Very High Risk (>6 points) disease according to the Revised International Prognostic Scoring System 2012 (IPSS-R).
* Clinical indication for treatment with azacitidine for MDS or AML.

Exclusion criteria:

* Patients with AML who are candidates for standard induction chemotherapy as first line treatment.
* Patients with known active CNS leukemia.
* Prior treatment with a smoothened inhibitor (SMOi) and/or hypomethylating agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (21):
  - University of Alabama at Birmingham the Kirklin Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook University Hospital Cancer Center, Stony Brook, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Einstein Center for Cancer, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Health System: Adult Bone Marrow Transplant Clinic, Durham, North Carolina
  - Duke University Health System, Duke University Hospital, Durham, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Investigational Chemotherapy Service, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance (SCCA), Seattle, Washington
  - University of Washington Medical Center (UWMC), Seattle, Washington
- Belgium (2):
  - Ziekenhuis Netwerk Antwerpen - Campus Stuivenberg, Antwerp
  - UZ Leuven, Leuven
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University Of Alberta Hospital, Edmonton, Alberta
- France (4):
  - CHU d'Amiens-Picardie - Hopital SUD, Amiens
  - Hopital Saint-Louis (AP-HP) - Service Hematologie Senior, Paris
  - Hospices Civils de Lyon - Hopital Lyon Sud- Hematologie, Pierre-Bénite
  - CHU de Tours-Hopital Bretonneau-Centre Regional de cancerologie Henry Kaplan, Tours
- Staedtisches Klinikum Braunschweig gGmbH, Braunschweig, Germany
- United Kingdom (3):
  - King's College Hospital, London
  - The Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sekeres MA, Schuster M, Joris M, Krauter J, Maertens J, Breems D, Gyan E, Kovacsovics T, Verma A, Vyas P, Wang ES, Ching K, O'Brien T, Gallo Stampino C, Ma WW, Kudla A, Chan G, Zeidan AM. A phase 1b study of glasdegib + azacitidine in patients with untreated acute myeloid leukemia and higher-risk myelodysplastic syndromes. Ann Hematol. 2022 Aug;101(8):1689-1701. doi: 10.1007/s00277-022-04853-4. Epub 2022 Apr 30. PMID 35488900
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371012&StudyName=A%20STUDY%20OF%20PF%2004449913%20IN%20COMBINATION%20WITH%20AZACITIDINE%20IN%20PATIENTS%20WITH%20PREVIOUSLY%20UNTREATED%20INTERMEDIATE%202%20OR%20HIGH%20RISK%20MYELODYSPLASTIC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants were enrolled and received combination therapy of glasdegib and azacitidine in the Lead-in Cohort (LIC). 31 participants were enrolled in the acute myeloid leukemia (AML) cohort, and 30 received glasdegib + azacitidine (1 participant withdrew consent before receiving treatment). 30 participants were enrolled and received glasdegib + azacitidine in the myelodysplastic syndrome (MDS) cohort.
Groups:
- Lead-in Cohort: Participants received subcutaneous (SC) administration of azacitidine daily at a dose of 75 mg/m2/day on Days 1-7 of every 28 days, and received oral self-administration of glasdegib daily and continuously at home with a starting dose of 100 mg once daily (QD). In Cycle 1 only, administration of glasdegib commenced on Day 2 of the cycle (C1D2) to permit drug-drug interaction (DDI) evaluation.
- AML Cohort: Participants received SC or intravenous (IV) administration of azacitidine at the starting dose of 75 mg/m2/day for 7 days every 28 days, and received oral self-administration of glasdegib daily and continuously at home with a starting dose of 100 mg QD.
- MDS Cohort: Participants received SC or IV administration of azacitidine at the starting dose of 75 mg/m2/day for 7 days every 28 days, and received oral self-administration of glasdegib daily and continuously at home with a starting dose of 100 mg QD.
Period: Overall Study
Arm/Group | Lead-in Cohort | AML Cohort | MDS Cohort
Started | 12 | 30 | 30
Completed | 0 | 0 | 0
Not Completed | 12 | 30 | 30
Not completed — Death | 8 | 24 | 17
Not completed — Lost to Follow-up | 1 | 3 | 1
Not completed — Other reason | 3 | 3 | 9
Not completed — Study Participation Terminated by Sponsor | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled and treated.
Groups:
- Lead-in Cohort: Participants received SC administration of azacitidine daily at a dose of 75 mg/m2/day on Days 1-7 of every 28 days, and received oral self-administration of glasdegib daily and continuously at home with a starting dose of 100 mg QD. In Cycle 1 only, administration of glasdegib commenced on Day 2 of the cycle (C1D2) to permit DDI evaluation.
- AML Cohort; MDS Cohort: Participants received SC or IV administration of azacitidine at the starting dose of 75 mg/m2/day for 7 days every 28 days, and received oral self-administration of glasdegib daily and continuously at home with a starting dose of 100 mg QD.
- Total: Total of all reporting groups
Arm/Group | Lead-in Cohort | AML Cohort | MDS Cohort | Total
Number analyzed (Participants) | 12 | 30 | 30 | 72
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0
  18-44 years | 0 | 0 | 0 | 0
  45-64 years | 3 | 3 | 7 | 13
  >=65 years | 9 | 27 | 23 | 59
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 7 | 16 | 22 | 45
  >=75 years | 5 | 14 | 8 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 6 | 23
  Male | 7 | 18 | 24 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 12 | 23 | 23 | 58
  Unknown or Not Reported | 0 | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 22 | 24 | 57
  Black or African American | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 0 | 2
  Other | 0 | 0 | 1 | 1
  Unknown | 0 | 6 | 5 | 11
  Not reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Lead-in Cohort (LIC)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. TEAEs were AEs that occurred after initiation of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator. Grades of AEs were defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE.
Time Frame: maximum of approximately 15 months
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
Participants
  All-causality TEAEs | 12
  Treatment-related TEAEs | 12
  Maximum Grade 3 or 4 TEAEs | 8

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) in the LIC
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: maximum of approximately 15 months
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
Participants
  All-causality SAEs | 9
  Treatment-related SAEs | 7

3. Primary Outcome: Number of Participants With Laboratory Abnormalities in the LIC
Description: Hematology lab parameters included activated partial thromboplastin time, hemoglobin, prothrombin international normalized ratio, lymphocyte, neutrophil, platelet, white blood cell; chemistry parameters included alanine aminotransferase, aspartate aminotransferase, alkaline aminotransferase, blood bilirubin, creatine phosphokinase, creatinine, calcium, blood glucose, potassium, magnesium, sodium, albumin, phosphate. Grades of lab abnormalities were defined by NCI CTCAE version 4.03. Grade 1(mild)=asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2(moderate)=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL;Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; disabling limiting self-care ADL;Grade 4=life-threatening consequences, urgent intervention indicated. Grade 1-4 results are reported.
Time Frame: maximum of approximately 16 months
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment. Number of participants analyzed = number of participants evaluable for this outcome measure (OM). Number analyzed = number of participants evaluable for this OM with at least 1 result of the specified laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 10
  Activated partial thromboplastin time prolonged | 5
  Anemia | 12
  Hemoglobin increased | 0
  international normalized ratio increased: number analyzed (Participants) | 11
  international normalized ratio increased | 8
  Lymphocyte count decreased | 9
  Lymphocyte count increased | 3
  Neutrophil count decreased | 10
  Platelet count decreased | 12
  White blood cell decreased | 11
  Alanine aminotransferase increased | 4
  Alkaline phosphatase increase | 0
  Aspartate aminotransferase increased | 2
  Blood bilirubin increased | 6
  creatine phosphokinase increased: number analyzed (Participants) | 11
  creatine phosphokinase increased | 0
  Creatinine increased | 11
  Hypercalcemia | 1
  Hyperglycemia | 1
  Hyperkalemia | 3
  Hypermagnesemia | 2
  Hypernatremia | 1
  Hypoalbuminemia | 5
  Hypocalcemia | 3
  Hypoglycemia | 1
  Hypokalemia | 3
  Hypomagnesemia | 2
  Hyponatremia | 6
  Hypophosphatemia | 4

4. Primary Outcome: Percentage of Participants Achieving Complete Remission (CR) in the AML and MDS Cohorts
Description: Percentage of participants achieving CR as defined by the 2017 European Leukemia Net (ELN) Response Criteria for all participants with AML and modified International Working Group (IWG) criteria (2006) for all participants with MDS in the expansion cohorts.
  For AML cohort, CR was defined as neutrophils ≥ 1 x 10^9/L, platelets ≥ 1 x 10^11/L, percentage of bone marrow blasts (BMB) <5% with no peripheral blasts and no blasts with Auer rods, no extramedullary disease (EMD), and transfusion independent.
  For MDS cohort, CR was defined as having responses of hemoglobin ≥11 g/dL, neutrophils ≥1 x 10^9/L, platelets ≥1 x 10^11/L, percentage of blasts = 0%, percentage of BMB≤5%, and normal maturation of all cell lines (note if has persistent dysplasia), and all responses must last at least 4 weeks.
Time Frame: maximum of 23 months in AML cohort and 34 months in MDS cohort
Population: The full analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- MDS Cohort: Participants received SC or IV administration of azacitidine with a starting dose of 75 mg/m2/day for 7 days every 28 days, and received daily oral administration of glasdegib at home with a starting dose of 100 mg QD.
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Percentage of participants | 20.0 [7.7 to 38.6] | 13.3 [3.8 to 30.7]

5. Secondary Outcome: Percentage of Participants Achieving Complete Remission (CR) + Partial Remission (PR) in the LIC
Description: Response rate (Percentage of participants achieving CR + PR among all the enrolled and treated patients) as defined by modified International Working Group (IWG) criteria (2006) in the LIC. CR was defined as having responses of hemoglobin ≥11 g/dL, neutrophils ≥1 x 10^9/L, platelets ≥1 x 10^11/L, percentage of blasts = 0%, percentage of BMB≤5%, and normal maturation of all cell lines (note if has persistent dysplasia), and all responses must last at least 4 weeks. PR was defined as meeting all CR criteria if abnormal before treatment except BMB, percentage of BMB decreased by ≥50% but still >5% for at least 4 weeks.
Time Frame: maximum of approximately 16 months
Population: The safety analysis population included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
Percentage of participants | 25.0

6. Secondary Outcome: Number of Participants With Efficacy Measures Other Than CR in the LIC
Description: Number of participants with efficacy measures other than CR as defined by modified IWG criteria (2006) in LIC, including marrow CR(mCR), stable disease(SD), hematologic improvement(HI). CR: hemoglobin≥11 g/dL, neutrophils≥1 x 10^9/L, platelets≥1 x 10^11/L, percentage of blasts=0%, percentage of BMB≤5%, normal maturation of all cell lines (note if has persistent dysplasia), all responses last at least 4 weeks. mCR: BMB≤5% & decreased by≥50%. SD: failure to achieve PR, no evidence of progression. HI: erythroid response (pretreatment<11g/dL): hemoglobin increase by≥1.5 g/dL, relevant reduction of units of red blood cell transfusions by at least 4 transfusions/8 weeks compared to pretreatment transfusion number in previous 8 weeks; platelet response (pretreatment<1x10^11/L): increase of≥30x10^9/L if starting with >20x10^9/L, and increase from <20x10^9/L to >20x10^9/L and by at least 100%; neutrophil response (pretreatment<1x10^9/L): at least a 100% increase, absolute increase >0.5x10^9/L
Time Frame: maximum of approximately 16 months
Population: The full analysis set was defined as all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
Participants
  marrow CR | 2
  stable disease | 4
  hematologic improvement of at least 1 lineage | 6

7. Secondary Outcome: Number of Participants With TEAEs in the AML and MDS Cohorts
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. TEAEs were AEs that occurred after initiation of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator. Grades of AEs were defined by NCI CTCAE version 4.03.Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE.
Time Frame: maximum of around 23 months in AML cohort and 40 months in MDS cohort
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Participants
  All-causality TEAEs | 30 | 30
  Treatment-related TEAEs | 29 | 29
  Maximum Grade 3 or 4 TEAEs | 20 | 25

8. Secondary Outcome: Number of Participants With SAEs in the AML and MDS Cohorts
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: maximum of around 23 months in AML cohort and 40 months in MDS cohort
Population: The safety analysis population included all participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Participants
  All-causality SAEs | 24 | 19
  Treatment-related SAEs | 8 | 9

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities in the AML and MDS Cohorts
Description: as for outcome 3
Time Frame: maximum of around 23 months in AML cohort and 40 months in MDS cohort
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment. Number of Participants Analyzed = number of participants evaluable for this outcome measure. Number Analyzed = number of participants with at least 1 observation of the given lab test.
Measure: Count of Participants; unit: Participants
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 2 | 2
  Activated partial thromboplastin time prolonged | 0 | 0
  Anemia: number analyzed (Participants) | 30 | 29
  Anemia | 30 | 29
  Hemoglobin increased: number analyzed (Participants) | 30 | 29
  Hemoglobin increased | 0 | 0
  international normalized ratio increased: number analyzed (Participants) | 2 | 2
  international normalized ratio increased | 0 | 2
  Leukocytosis: number analyzed (Participants) | 30 | 29
  Leukocytosis | 0 | 1
  Lymphocyte count decreased: number analyzed (Participants) | 30 | 27
  Lymphocyte count decreased | 23 | 24
  Lymphocyte count increased: number analyzed (Participants) | 30 | 27
  Lymphocyte count increased | 6 | 2
  Neutrophil count decreased: number analyzed (Participants) | 30 | 28
  Neutrophil count decreased | 25 | 25
  Platelet count decreased: number analyzed (Participants) | 30 | 29
  Platelet count decreased | 29 | 26
  White blood cell decreased: number analyzed (Participants) | 30 | 29
  White blood cell decreased | 22 | 27
  Alanine aminotransferase increased: number analyzed (Participants) | 30 | 29
  Alanine aminotransferase increased | 13 | 12
  Alkaline phosphatase increased: number analyzed (Participants) | 30 | 29
  Alkaline phosphatase increased | 7 | 8
  Aspartate aminotransferase increased: number analyzed (Participants) | 30 | 29
  Aspartate aminotransferase increased | 11 | 9
  Blood bilirubin increased: number analyzed (Participants) | 30 | 29
  Blood bilirubin increased | 3 | 10
  creatine phosphokinase increased: number analyzed (Participants) | 29 | 28
  creatine phosphokinase increased | 5 | 4
  creatinine increased: number analyzed (Participants) | 30 | 29
  creatinine increased | 29 | 28
  Hypercalcemia: number analyzed (Participants) | 30 | 29
  Hypercalcemia | 3 | 0
  Hyperglycemia: number analyzed (Participants) | 30 | 29
  Hyperglycemia | 3 | 4
  Hyperkalemia: number analyzed (Participants) | 30 | 29
  Hyperkalemia | 6 | 6
  Hypermagnesemia: number analyzed (Participants) | 30 | 29
  Hypermagnesemia | 1 | 2
  Hypernatremia: number analyzed (Participants) | 30 | 29
  Hypernatremia | 2 | 1
  Hypoalbuminemia: number analyzed (Participants) | 30 | 29
  Hypoalbuminemia | 22 | 19
  Hypocalcemia: number analyzed (Participants) | 30 | 29
  Hypocalcemia | 3 | 11
  Hypoglycemia: number analyzed (Participants) | 30 | 29
  Hypoglycemia | 4 | 3
  Hypokalemia: number analyzed (Participants) | 30 | 29
  Hypokalemia | 8 | 3
  Hypomagnesemia: number analyzed (Participants) | 30 | 29
  Hypomagnesemia | 12 | 10
  Hyponatremia: number analyzed (Participants) | 30 | 29
  Hyponatremia | 18 | 12
  Hypophosphatemia: number analyzed (Participants) | 30 | 29
  Hypophosphatemia | 13 | 7

10. Secondary Outcome: Number of Participants With Disease-Specific Efficacy Measures in the AML Cohort
Description: Number of participants with partial hematologic recovery (CRh), CR with incomplete blood count recovery (CRi), partial remission (PR), stable disease (SD), and morphologic leukemia free state (MLFS). CRh: neutrophils>5x10^8/L, platelets>5x10^10/L, BMB<5%, no peripheral blasts, no blasts with Auer rods, no extramedullary disease (EMD), not qualifying for CR. CRi: neutrophils <1x10^9/L or platelets<1x10^11/L; BMB <5%, no peripheral blasts, no blasts with Auer rods; no EMD; neutrophils or platelets not recovered; not qualifying for CRh. PR: neutrophils ≥1x10^9/L; platelets ≥1x10^11/L; blasts decreased to 5-25% and ≥50% decrease from pretreatment; blasts≤5% if Auer rod positive. SD: ≥3 months of absence of CR without minimal residual disease (CRMRD-), CR, CRh, CRi, PR, and MLFS, criteria for PD not met. MLFS: neutrophils <1x10^9/L and platelets<1x10^11/L, BMB<5%, no blasts with Auer rods; no EMD; neutrophils and platelets not recovered; not qualifying for CRi
Time Frame: maximum of 23 months
Population: The full analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AML Cohort
Number analyzed (Participants) | 30
Participants
  partial hematologic recovery (CRh) | 0
  CR with incomplete blood count recovery (CRi) | 1
  partial remission (PR) | 2
  morphologic leukemia free state (MLFS) | 1
  stable disease (SD) | 6

11. Secondary Outcome: Number of Participants With Disease-Specific Efficacy Measures in the MDS Cohort
Description: Number of participants with PR, mCR, SD, complete or partial cytogenetic response, and HI. PR: BMB >5% and decreased by ≥50% (at least 4 weeks), meeting all CR criteria if abnormal before treatment except BMB. mCR: BMB ≤5% and decreased by ≥50%. SD: failure to achieve PR, no evidence of progression. Complete or partial cytogenic response: disappearance of chromosomal abnormality without new ones, or ≥ 50% reduction of chromosomal abnormality. HI: erythroid response (pretreatment <11g/dL): hemoglobin increase by≥1.5 g/dL, relevant reduction of units of red blood cell transfusions by at least 4 transfusions/8 weeks compared to pretreatment transfusion number in previous 8 weeks; platelet response (pretreatment <1x10^11/L): increase of ≥30x10^9/L if starting with >20x10^9/L, and increase from <20x10^9/L to >20x10^9/L and by at least 100%; neutrophil response (pretreatment <1x10^9/L): at least a 100% increase, absolute increase >0.5x10^9/L.
Time Frame: maximum of 34 months
Population: The full analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MDS Cohort
Number analyzed (Participants) | 30
Participants
  PR | 3
  mCR | 5
  SD | 8
  Complete cytogenetic response | 5
  Partial cytogenetic response | 1
  HI of at least 1 lineage | 9
  HI of at least 1 lineage without CR or PR | 3

12. Secondary Outcome: Kaplan-Meier Estimate of Median Overall Survival (OS) in the AML and MDS Cohorts
Description: Overall survival (OS) was defined as the time from date of first study treatment to date of death from any cause. Patients last known to be alive were to be censored at the date of last contact. OS was analyzed and displayed graphically for each expansion cohort separately using the Kaplan-Meier method. The median event time and corresponding two-sided 95%CI were provided for each cohort. OS was first analyzed when the primary endpoint of CR was analyzed in the respective expansion cohort.
Time Frame: maximum of approximately 32 months in AML cohort and 32 months in MDS cohort
Population: The full analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Months | 9.2 [6.2 to 14.0] | 17.8 [9.3 to NA] — The upper limit was not estimable due to insufficient number of participants with events.

13. Secondary Outcome: Duration of CR in the AML and MDS Cohorts
Description: Duration of CR was defined as the duration from date of first achieving CR to the date of disease progression (relapse) after CR, or death due to any cause. Participants last known to be alive who were free from disease progression or relapse after CR were censored at the date of the last assessment that verified their disease status. Duration of CR was analyzed using the Kaplan-Meier method. Disease progression was defined as: percentage of bone marrow blasts increased by ≥50% to >5% (for participants with <5% blasts at screening), >10% (for participants with 5-10% blasts at screening), >20% (for participants with 11-20% blasts at screening) or >30% (for participants with 21-30% blasts at screening), and with any of the following condition: at least 50% decrease from maximum remission/response in granulocytes or platelets; reduction in hemoglobin by ≥2 g/dL; transfusion dependence.
Time Frame: maximum of 23 months in AML cohort and 34 months in MDS cohort
Population: The analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Median (Full Range); unit: Months
Groups:
- AML Cohort; MDS Cohort: Participants received SC or IV administration of azacitidine with a starting dose of 75 mg/m2/day for 7 days every 28 days, and received daily oral administration of glasdegib at home with a starting dose of 100 mg QD.
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Months | 5.78 [0.03 to 16.85] | 6.18 [0.72 to 18.07]

14. Secondary Outcome: Time to CR in the AML and MDS Cohorts
Description: Time to CR was defined for participants in the expansion cohorts who had achieved response on study as the time from date of the first dose of study drug to date of the first documentation of response. Time to CR was analyzed using the Kaplan-Meier method.
Time Frame: maximum of 23 months in AML cohort and 34 months in MDS cohort
Population: The analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
Months | 5.54 [3.12 to 5.98] | 4.39 [3.71 to 5.55]

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Glasdegib Dosed in Combination With Azacitidine (C1D7) and When Dosed Alone (C1D15) in the Lead-in Cohort
Description: Maximum plasma concentration of glasdegib dosed in combination with azacitidine (C1D7) and when dosed alone (C1D15) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: Pre-dose and 0.25, 1, 4, 6, 24 hours post-dose on Cycle 1 Day 7 and Cycle 1 Day 15
Population: The PK concentration analysis set included all participants who received treatment and had at least 1 value of analyte concentration of glasdegib or azacitidine available. Number of participants analyzed = number of participants evaluable for this OM. Number analyzed = number of participants with evaluable results at the specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL)
  C1D7 | 1013 (58)
  C1D15: number analyzed (Participants) | 9
  C1D15 | 991.4 (57)

16. Secondary Outcome: Area Under the Plasma Concentration Curve From Time Zero to End of Dosing Interval (AUCtau) of Glasdegib Dosed in Combination With Azacitidine (C1D7) and When Dosed Alone (C1D15) in the Lead-in Cohort
Description: Area under the plasma concentration curve from time zero to end of dosing interval (AUCtau) of glasdegib dosed in combination with azacitidine (C1D7) and when dosed alone (C1D15) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: Pre-dose and 0.25, 1, 4, 6, 24 hours post-dose on Cycle 1 Day 7 and Cycle 1 Day 15
Population: The PK parameter analysis set included all participants who received study treatment and had at least 1 of the PK parameters of interest. Number of participants analyzed = number of participants evaluable for this OM. Number analyzed = number of participants with evaluable results at the specific timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour/milliliter (ng*hr/mL)
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
nanogram * hour/milliliter (ng*hr/mL)
  C1D7 | 13230 (49)
  C1D15: number analyzed (Participants) | 9
  C1D15 | 14350 (61)

17. Secondary Outcome: Time to First Occurrence of Maximum Plasma Concentration (Tmax) of Glasdegib Dosed in Combination With Azacitidine (C1D7) and When Dosed Alone (C1D15) in the Lead-in Cohort
Description: Time to first occurrence of maximum plasma concentration of glasdegib dosed in combination with azacitidine (C1D7) and when dosed alone (C1D15) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: Pre-dose and 0.25, 1, 4, 6, 24 hours post-dose on Cycle 1 Day 7 and Cycle 1 Day 15
Population: as for outcome 16
Measure: Median (Full Range); unit: hour
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
hour
  C1D7 | 1.050 [1.00 to 5.70]
  C1D15: number analyzed (Participants) | 9
  C1D15 | 1.500 [1.00 to 6.02]

18. Secondary Outcome: Cmax of Azacitidine Dosed in Combination With Glasdegib (C1D7) and When Dosed Alone (C1D1) in the Lead-in Cohort
Description: Maximum plasma concentration of azacitidine dosed in combination with glasdegib (C1D7) and when dosed alone (C1D1) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: 0.25, 0.5, 1, 2, 6 hours post-dose on Cycle 1 Day 1, predose and 0.25, 0.5, 1, 2, 6 hours postdose on Cycle 1 Day 7
Population: The PK concentration analysis set included all participants who received treatment and had at least 1 value of analyte concentration of glasdegib or azacitidine available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
ng/mL
  C1D1 | 778.5 (23)
  C1D7 | 716.9 (32)

19. Secondary Outcome: Area Under the Plasma Concentration Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Azacitidine Dosed in Combination With Glasdegib (C1D7) and When Dosed Alone (C1D1) in the Lead-in Cohort
Description: Area under the plasma concentration curve from time zero to extrapolated infinite time of azacitidine dosed in combination with glasdegib (C1D7) and when dosed alone (C1D1) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: 0.25, 0.5, 1, 2, 6 hours post-dose on Cycle 1 Day 1, predose and 0.25, 0.5, 1, 2, 6 hours postdose on Cycle 1 Day 7
Population: The PK parameter analysis set included all participants who received study treatment and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
ng*hr/mL
  C1D1 | 1319 (19)
  C1D7 | 1260 (21)

20. Secondary Outcome: Tmax of Azacitidine Dosed in Combination With Glasdegib (C1D7) and When Dosed Alone (C1D1) in the Lead-in Cohort
Description: Time to first occurrence of maximum plasma concentration of azacitidine dosed in combination with glasdegib (C1D7) and when dosed alone (C1D1) in the Lead-in Cohort was estimated using non-compartmental analysis.
Time Frame: 0.25, 0.5, 1, 2, 6 hours post-dose on Cycle 1 Day 1, predose and 0.25, 0.5, 1, 2, 6 hours postdose on Cycle 1 Day 7
Population: as for outcome 19
Measure: Median (Full Range); unit: hour
Arm/Group | Lead-in Cohort
Number analyzed (Participants) | 12
hour
  C1D1 | 0.5000 [0.000 to 1.00]
  C1D7 | 0.5000 [0.250 to 1.08]

21. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Glasdegib on Cycle 1 Day 15 and Cycle 2 Day 1 in the AML and MDS Cohorts
Description: Trough plasma concentration was defined as the estimated lowest concentration before next dose administration.
Time Frame: Pre-dose and 1 and 4 hours post-dose on Cycle 1 Day 15 (C1D15) and Cycle 2 Day 1 (C2D1)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AML Cohort | MDS Cohort
Number analyzed (Participants) | 30 | 30
ng/mL
  C1D15: number analyzed (Participants) | 25 | 22
  C1D15 | 468.440 (88) | 308.144 (95)
  C2D1: number analyzed (Participants) | 17 | 18
  C2D1 | 462.806 (110) | 167.483 (52)

22. Secondary Outcome: Number of Participants Meeting Categorical Criteria of QTcF Values in LIC, AML and MDS Cohorts
Description: Number of participants that met categorical criteria of QTcF values in LIC, AML and MDS cohorts
Time Frame: maximum of approximately 15 months in the LIC cohort, 23 months in AML cohort, and 40 months in MDS cohort
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort | AML Cohort | MDS Cohort
Number analyzed (Participants) | 12 | 30 | 30
Participants
  Maximum QTcF interval <450 ms | 5 | 16 | 17
  450 ms <=Maximum QTcF interval <480 ms | 2 | 6 | 7
  480 ms <=Maximum QTcF interval <500 ms | 4 | 5 | 4
  Maximum QTcF interval ≥500 ms | 1 | 3 | 2
  QTcF maximum increase from baseline <30 ms | 3 | 18 | 21
  30 ms <= QTcF maximum increase from baseline <60 ms | 7 | 10 | 7
  QTcF maximum increase from baseline >=60 ms | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: maximum of approximately 15 months in the LIC cohort, 23 months in the AML cohort, and 40 months in the MDS cohort
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Lead-in Cohort | AML Cohort | MDS Cohort
All-Cause Mortality (participants affected / at risk) | 9/12 | 25/30 | 17/30
Serious Adverse Events (participants affected / at risk) | 9/12 | 24/30 | 19/30
Other Adverse Events (participants affected / at risk) | 12/12 | 29/30 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Cohort (N=12) | AML Cohort (N=30) | MDS Cohort (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 3 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
General physical health deterioration (General disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 5
Septic shock (Infections and infestations) | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 4 | 2
Urosepsis (Infections and infestations) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 2 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 — Investigator entry: unexpected death (reason of death unknown)
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Cohort (N=12) | AML Cohort (N=30) | MDS Cohort (N=30)
Anaemia (Blood and lymphatic system disorders) | 9 | 6 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2
Asthenia (General disorders) | 2 | 3 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 16 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 9 | 18 | 15
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 16 | 14
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 4 | 2
Nausea (Gastrointestinal disorders) | 8 | 19 | 21
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral dysaethesia (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 13 | 10
Chest pain (General disorders) | 0 | 2 | 0
Chills (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 6 | 8 | 9
General physical health deterioration (General disorders) | 0 | 2 | 0
Injection site erythema (General disorders) | 3 | 2 | 0
Injection site irritation (General disorders) | 1 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 3 | 0
Injection site reaction (General disorders) | 2 | 2 | 6
Oedema peripheral (General disorders) | 3 | 4 | 9
Pain (General disorders) | 1 | 5 | 2
Pyrexia (General disorders) | 2 | 8 | 4
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 4 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 2
Sepsis (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 8 | 7
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increase (Investigations) | 0 | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 2
Blood bilirubin increased (Investigations) | 2 | 3 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 4 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 5 | 5 | 3
Heart rate irregular (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 3 | 2
Lymphocyte count decreased (Investigations) | 0 | 4 | 4
Neutrophil count decreased (Investigations) | 0 | 2 | 11
Platelet count decreased (Investigations) | 0 | 5 | 11
Weight decreased (Investigations) | 5 | 5 | 6
White blood cell count decreased (Investigations) | 1 | 7 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 7 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 9 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 3 | 7
Dizziness postural (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 5 | 4 | 13
Headache (Nervous system disorders) | 0 | 3 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 3
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 4 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0
Taste disorder (Nervous system disorders) | 1 | 3 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 6 | 6
Mental status change (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 3 | 3
Dysuria (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 2 | 3 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0
Hypotension (Vascular disorders) | 2 | 3 | 7
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Serum ferritin decreased (Investigations) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02367456/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02367456/SAP_001.pdf